CLINICAL TRIAL: NCT01963507
Title: Effects of a Resistance Training Period on Blood Pressure of Hypertensive Elderlies: Influence of the Polymorphism of the Angiotensin Converting Enzyme
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Federal University of São Paulo (Other)
Collaborators: Fundação de Amparo à Pesquisa do Estado de São Paulo (Other Government)
Responsible Party: Principal Investigator, Alessandra Medeiros, PhD, Federal University of São Paulo
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ACE RT
Record Dates: First submitted 2013-10-09; First posted 2013-10-16 (Estimated); Last update posted 2013-10-16 (Estimated); Status verified 2013-10

CONDITIONS: Hypertension
MeSH Terms: conditions — Hypertension | interventions — Resistance Training

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Resistance training (Experimental): Resistance training performed three times at week for 16 weeks, in 8 exercises for the main muscles, the protocol of 3 sets of 10 repetitions with intensity of 50% of 1 maximum repetition (MR).
  Interventions: Behavioral: Resistance training
- Control (No Intervention)

INTERVENTIONS:
Behavioral: Resistance training — Resistance training performed three times at week for 16 weeks, in 8 exercises for the main muscles, the protocol of 3 sets of 10 repetitions with intensity of 50% of 1 maximum repetition (MR).
  Arms: Resistance training

SUMMARY:
The study aimed to evaluate the chronic effects of resistance training on blood pressure and biochemical exams in hypertensive elderlies and the influence of the polymorphism of the angiotensin converting enzyme in these response.

DETAILED DESCRIPTION:
To investigate the chronic effects of resistance training on blood pressure and biochemical exams in elderly, 135 hypertensive elderlies were divided into 2 groups: trained and control. The trained group was submitted to a resistance training period. Before the 16 weeks ACE gene was genotyped (PCR). Before and after 16 weeks, blood pressure (ambulatory), HDL-cholesterol, Total cholesterol, Glycemia, Triacylglycerol (colorimetric assay) and plasminogen activator inhibition (PAI-1), intercellular adhesion molecule (ICAM-1), vascular endothelial cell adhesion molecule (VCAM-1), Adiponectin, tumor necrosis factor alpha (TNF-alpha), C Reactive Protein, Angiotensin II, Angiotensin Converting Enzyme, Angiotensin 1-7, (ELISA assay) were measured.

ELIGIBILITY:
Inclusion Criteria:

* Hypertensives
* Age 60 to 85 years
* Nonactive

Exclusion Criteria:

* Orthopedic problems or other problem that prevented the exercises
* Change in drug treatment during protocol
* Absence in more than 25% of the exercise sessions

Ages: 60 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 136 (Actual)
Dates: Start 2010-04; Primary Completion 2013-04 (Actual); Study Completion 2013-04 (Actual)

PRIMARY OUTCOMES:
Blood Pressure | 16 weeks
  Blood pressure was measured by Ambulatorial Monitoring Blood Pressure before and after 16 weeks of intervention.

SECONDARY OUTCOMES:
HDL-cholesterol | 16 weeks
  HDL-cholesterol was analyzed by colorimetric assay, before and after 16 weeks of intervention.
Total Cholesterol | 16 weeks
  Total cholesterol was analyzed by colorimetric assay, before and after 16 weeks of intervention.
Glycemia | 16 weeks
  Glycemia was analyzed by colorimetric assay, before and after 16 weeks of intervention.
Triacylglycerol | 16 weeks
  Triacylglycerol was analyzed by colorimetric assay, before and after 16 weeks of intervention.
PAI-1 | 16 weeks
  PAI-1 was analyzed by ELISA assay, before and after 16 weeks of intervention.
ICAM-1 | 16 weeks
  ICAM-1 was analyzed by ELISA assay, before and after 16 weeks of intervention.
VCAM-1 | 16 weeks
  VCAM-1 was analyzed by ELISA assay, before and after 16 weeks of intervention.
Adiponectin | 16 weeks
  Adiponectin was analyzed by ELISA assay, before and after 16 weeks of intervention.
TNF alpha | 16 weeks
  TNF alpha was analyzed by ELISA assay, before and after 16 weeks of intervention.
C Reactive Protein | 16 weeks
  C Reactive Protein was analyzed by ELISA assay, before and after 16 weeks of intervention.
Angiotensin II | 16 weeks
  Angiotensin II was analyzed by ELISA assay, before and after 16 weeks of intervention.
Angiotensin Converting Enzyme | 16 weeks
  Angiotensin Converting Enzyme was analyzed by ELISA assay, before and after 16 weeks of intervention.
Angiotensin 1-7 | 16 weeks
  Angiotensin 1-7 was analyzed by ELISA assay, before and after 16 weeks of intervention.

CONTACTS AND LOCATIONS:
Locations (1):
- UNIMED, Santos, São Paulo, Brazil